CLINICAL TRIAL: NCT00848536
Title: A Multi-Center, Double-Masked Study of the Safety and Efficacy of Travoprost APS Compared to TRAVATAN® in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Efficacy Study of Travoprost APS Versus TRAVATAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-08-40; 2008-006027-31 (EudraCT Number)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Ophthalmic Solutions; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRAVATAN APS (Experimental): One drop once daily in the evening for 3 months
  Interventions: Drug: Travoprost 0.004% (POLYQUAD-preserved) Eye Drops, Solution
- TRAVATAN (Active Comparator): One drop once daily in the evening for 3 months
  Interventions: Drug: Travoprost 0.004% (BAK-preserved) Eye Drops, Solution

INTERVENTIONS:
Drug: Travoprost 0.004% (POLYQUAD-preserved) Eye Drops, Solution — One drop once daily in the evening for 3 months
  Arms: TRAVATAN APS
Drug: Travoprost 0.004% (BAK-preserved) Eye Drops, Solution — One drop once daily in the evening for 3 months
  Arms: TRAVATAN

SUMMARY:
A Multi-Center Double-masked Study of the Safety and Efficacy of Travoprost APS Compared to TRAVATAN in Patients with Open-angle Glaucoma or Ocular Hypertension

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, either gender and any race.
* Open Angle Glaucoma (OAG) or Ocular Hypertension (OHT).
* Not currently on any IOP-lowering medication or currently on a stable treatment (i.e, at least 30 days) with and IOP-lowering monotherapy.
* All patients: Mean IOP in same eye (at both Eligibility 1 & 2 Visits):

  ≥ 24 and ≤ 36 mmHg at 9 AM; and ≥ 21 and ≤ 36 mmHg at 11 AM & 4 PM.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential not meeting conditions set in the protocol.
* Severe central visual field loss.
* Angle Shaffer grade < 2.
* Cup/disc ratio > 0.8 (horizontal or vertical measurement).
* Best corrected visual acuity (VA) score worse than 55 ETDRS letters read (equivalent to approximately 20/80 Snellen or 0.25 decimal).
* Intraocular surgery or trauma within last 6 months.
* Any abnormality preventing reliable applanation tonometry.
* History of or current ocular pathology (including severe dry eye) that would affect the conduct of the study.
* Allergy/hypersensitivity to study medications.
* Unable to discontinue use of all IOP-lowering medications for a minimum wash-out period of 5 to 28 days prior to the Eligibility Visit.
* Less than 30 days stable dosing regimen of medications used on a chronic basis that may affect IOP.
* Use of any additional topical or systemic ocular hypotensive medication during the study.
* Therapy with another investigational agent within 30 days prior to the Screening visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 30 study centers: 8 in the US, 6 in Mexico, 2 in Brazil, 4 in India, 2 in Australia, 2 in New Zealand, 2 in Latvia, and a single site in each: Taiwan, France, Belgium, and Italy.
Period: Overall Study
Arm/Group | TRAVATAN APS | TRAVATAN
Started | 185 | 186
Completed | 181 | 179
Not Completed | 4 | 7
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Noncompliance | 1 | 0
Not completed — Inadequate Control of IOP | 1 | 1
Not completed — Patient Moved | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRAVATAN APS | TRAVATAN | Total
Number analyzed (Participants) | 185 | 186 | 371
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 109 | 203
  >=65 years | 91 | 77 | 168
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 115 | 227
  Male | 73 | 71 | 144

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure at 9:00 am
Description: For an individual patient, two consecutive IOP measurements for each eye were taken. The mean IOP values for each individual patient's eye were rounded up to the next whole number if the value was ≥ 0.5 mmHg
  All IOP measurements were performed with a Goldmann applanation tonometer. All IOP measurements for any individual subject were to be performed preferably by the same operator using the same tonometer.
  Mean IOP for the patient's worse eye at baseline was used in the primary endpoint analysis. If both eyes were equal, then the right eye was selected for analysis
Time Frame: 3 months (measured at 9:00 am)
Population: Per-Protocol. Patients who received study medication, satisfied pre-randomization criteria and satisfied protocol criteria at the specific time point were considered evaluable for PP analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | TRAVATAN APS | TRAVATAN
Number analyzed (Participants) | 172 | 172
mmHg | 17.9 (0.25) | 18.1 (0.25)
Statistical Analysis 1: Comparison: TRAVATAN APS vs TRAVATAN; A hypothesis test was performed using a repeated measures analysis of variance model. For the test of non-inferiority, a two-sided 95% confidence intervals for the treatment group difference in mean IOP at each visit and time point was constructed based on analysis of variance; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 1.5 mmHg; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.35 — Treatment group differences were calculated as the mean IOP in the Travoprost APS group minus the mean IOP in the Travatan group. Non-inferiority was demonstrated if the upper 95% CL of the between treatment difference in mean IOP was < 1.5 mmHg

2. Primary Outcome: Mean Intraocular Pressure at 11:00 am
Description: as for outcome 1
Time Frame: 3 months (measured at 11:00 am)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | TRAVATAN APS | TRAVATAN
Number analyzed (Participants) | 171 | 171
mmHg | 17.4 (0.25) | 17.5 (0.25)
Statistical Analysis 1: Comparison: TRAVATAN APS vs TRAVATAN; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 1.5 mmHg; Median Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 00.6], Standard Error of Mean 0.35 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Intraocular Pressure at 4:00 pm
Description: as for outcome 1
Time Frame: 3 months (measured at 4:00 pm)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | TRAVATAN APS | TRAVATAN
Number analyzed (Participants) | 171 | 171
mmHg | 16.9 (0.25) | 17.1 (0.25)
Statistical Analysis 1: Comparison: TRAVATAN APS vs TRAVATAN; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 1.5 mmHg; Median Difference (Final Values) = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.35 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | TRAVATAN APS | TRAVATAN
Serious Adverse Events (participants affected / at risk) | 1/185 | 2/186
Other Adverse Events (participants affected / at risk) | 32/185 | 35/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRAVATAN APS (N=185) | TRAVATAN (N=186)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRAVATAN APS (N=185) | TRAVATAN (N=186)
Ocular hyperaemia (Eye disorders) | 21 (22) | 19 (22)
Eye irritation (Eye disorders) | 7 (8) | 11 (12)
Conjunctival hyperaemia (Eye disorders) | 8 (9) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less